CLINICAL TRIAL: NCT05727540
Title: The Cohort Study of Uveitis Patients Based on Real-world Data
Brief Title: The Cohort Study of Uveitis Patients
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ227
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-06

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Noninfectious uveitis
- Infectious uveitis

SUMMARY:
This study intends to explore the epidemiology, pathogenesis, clinical manifestations, diagnosis and treatment of uveitis. This is a cohort study. The outcome of the study is the activity of inflammation and visual prognosis. The purpose of this study is to determine the optimal diagnosis and treatment scheme for uveitis patients based on real-world data.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis is uveitis; The agreement of enrolling this study;

Exclusion Criteria:

* Uveitis during the first month after any intraocular surgery; <18 years; pregnant and lactating women; other conditions are unsuitable for participation in this study by the investigator such as mental abnormalities.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are adult uveitis patients.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 12 months post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The range of inflammatory chorioretinal and/or inflammatory retinal vascular lesions | 12 months post-treatment
  inflammatory chorioretinal and/or inflammatory retinal vascular lesions were evaluated by fundus fluorescein angiography and indocyanine green angiography

SECONDARY OUTCOMES:
Best corrected visual acuity | 1 month post-treatment
  Best corrected visual acuity
Best corrected visual acuity | 3 months post-treatment
  Best corrected visual acuity
Best corrected visual acuity | 6 months post-treatment
  Best corrected visual acuity
Best corrected visual acuity | 12 months post-treatment
  Best corrected visual acuity
Best corrected visual acuity | 24 months post-treatment
  Best corrected visual acuity
Best corrected visual acuity | 36 months post-treatment
  Best corrected visual acuity
The number of intraocular pressure | 1 month post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
The number of intraocular pressure | 3 months post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
The number of intraocular pressure | 6 months post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
The number of Intraocular pressure | 12 months post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
The number of Intraocular pressure | 24 months post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
The number of Intraocular pressure | 36 months post-treatment
  The number of Intraocular pressure was examed by non-contact tonometer
Central retinal thickness | 1 month post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
Central retinal thickness | 3 months post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
Central retinal thickness | 6 months post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
Central retinal thickness | 12 months post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
Central retinal thickness | 24 months post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
Central retinal thickness | 36 months post-treatment
  Central retinal thickness was evaluated by Optical Coherence Tomography
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 1 month post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 3 months post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 6 months post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 24 months post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The socre of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system | 36 months post-treatment
  activity of anterior chamber inflammation based on the Standardization of Uveitis Nomenclature (SUN) scoring system
The range of inflammatory chorioretinal and/or inflammatory retinal vascular lesions | 3 months post-treatment
  inflammatory chorioretinal and/or inflammatory retinal vascular lesions were evaluated by fundus fluorescein angiography and indocyanine green angiography
The range of inflammatory chorioretinal and/or inflammatory retinal vascular lesions | 6 months post-treatment
  inflammatory chorioretinal and/or inflammatory retinal vascular lesions were evaluated by fundus fluorescein angiography and indocyanine green angiography
The range of inflammatory chorioretinal and/or inflammatory retinal vascular lesions | 24 months post-treatment
  inflammatory chorioretinal and/or inflammatory retinal vascular lesions were evaluated by fundus fluorescein angiography and indocyanine green angiography
The range of inflammatory chorioretinal and/or inflammatory retinal vascular lesions | 36 months post-treatment
  inflammatory chorioretinal and/or inflammatory retinal vascular lesions were evaluated by fundus fluorescein angiography and indocyanine green angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China